CLINICAL TRIAL: NCT06693570
Title: A Randomized Controlled Multicenter Clinical Trial Evaluating Intact Fish Skin Graft and Standard of Care Versus Standard of Care Alone in Nonhealing Venous Leg Ulcers
Brief Title: Evaluating Intact Fish Skin Graft and Standard of Care Versus Standard of Care Alone in Nonhealing Venous Leg Ulcers
Acronym: THOR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS-1010; Pro00081893 (Other: Advarra IRB)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Venous Leg Ulcer (VLU); Venous Leg Ulcers; Venous Leg; Nonhealing Venous Leg Ulcer
Keywords: Fish Skin Graft; Intact Fish Skin Graft
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Multicenter Prospective Randomized Comparative Effectiveness Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intact Fish Skin Graft (IFSG) + Standard of Care (Experimental): Up to 12 visits with Intact Fish Skin Graft (IFSG) + Standard of Care.
  Interventions: Other: Intact Fish Skin Graft (IFSG) + Standard of Care
- Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Intact Fish Skin Graft (IFSG) + Standard of Care — Participants will receive weekly applications of MariGen and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Intact Fish Skin Graft (IFSG) + Standard of Care
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine the between-arm difference in the proportion of subjects achieving complete closure of hard-to-heal venous leg ulcers (VLU) between Intact Fish Skin Graft plus standard of care (IFSG/SOC) versus standard of care alone (SOC) over 12 weeks.

DETAILED DESCRIPTION:
This is a randomized controlled multicenter clinical trial evaluating intact fish skin grand and standard of care vs. standard of care alone in nonhealing venous leg ulcers. The product classifies as a medical device and consists of a full thickness fish-skin that has been processed using Kerecis™ Limited's proprietary EnviroIntact™ method.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a nonhealing venous leg ulcer present for a minimum of 4 weeks and cannot have received more than 52 weeks of high-level compression prior to the initial screening visit.
3. No visible signs of healing objectively, less than 40% reduction in wound size in the last 4 weeks.
4. At randomization, subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 25 cm2 measured post-debridement.
5. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
6. If the potential subject has two or more ulcers, and they are separated by at least 2 cm post-debridement, the largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer. If the potential subject has two or more ulcers and they are separated by less than 2cm, the entire wound area is designated as the target ulcer.
7. Subjects must have a Functional Ambulatory Category Score (FACS) of 3 or greater.
8. Subjects must consent to using the prescribed compression method for the duration of the study.
9. Subjects must agree to attend the weekly study visits required by the protocol.
10. Subjects must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The index ulcer is determined to be due to a condition other than venous insufficiency.
3. The target ulcer exposes muscle, tendon, or bone.
4. The target ulcer exhibits overt clinical signs and symptoms of infection with cellulitis surrounding the wound margin.
5. The target ulcer has known or suspected skin malignancy.
6. The target ulcer has been previously exposed to radiation.
7. The target ulcer duration is greater than one year having received high level compression without closure for a year or more.
8. The potential subject has end stage renal disease requiring dialysis.
9. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
10. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
11. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a cellular or tissue-based product (CTP) in the 30 days prior to the initial screening visit.
12. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
13. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
14. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Digital planimetry is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
15. The surface area measurement of the target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
16. The potential subject has a Functional Ambulatory Category Score (FACS) of less than 3.
17. The potential subject has a body mass index (BMI) greater than 42
18. In the last 8 weeks the patient has undergone revascularization (surgical or stenting) to the affected leg.
19. Venous intervention in the affected limb in the last 30 days.
20. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator.
21. Pregnancy at enrollment or women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
22. Know allergy to any of the components of fish skin or bovine collagen.
23. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
24. A subject with a disorder that would create unacceptable risk of post-operative complications is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of target ulcers achieving complete wound closure | [Time Frame: 1-12 Weeks]
  The percentage of target ulcers achieving complete wound closure in 12 weeks

SECONDARY OUTCOMES:
Time to closure | [Time Frame: 1-12 weeks]
  The time to closure of the target ulcers over 12 weeks.
Percent area change | [Time Frame: 1-12 weeks]
  Percentage wound area change from TV-1 to TV-13 measured weekly with digital photographic planimetry and physical examination.
Adverse Events | [Time Frame: 1-12 weeks]
  The number of adverse events.
Change in pain in target ulcer | [Time Frame: 1-12 weeks]
  Change in pain in the target ulcer assessed using the Visual Analog Scale VAS scale from TV-1 to TV-13
Visits and product applications needed to close the ulcer | [Time Frame: 1-12 weeks]
  The number of visits and product applications needed to close the ulcer
Quality of life using the Wound quality of Life questionare wQOL | [Time Frame: 1-12 weeks]
  Change in quality of life using the wQOL checklist [TV-1, TV-4, TV-8, and TV-12/Final Visit].
Determine improvement in Quality of Life - Forgotten Wound Score FWS | [Time Frame: 1-12 weeks]
  Quality of Life assessed using the Forgotten Wound Score. The scale has a score of 0 to 100- 100 being the worst outcome meaning the wound bothers the subject most of the time. [TV-1, TV-4, TV-8, and TV-12/Final Visit].

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Group- Monroeville, Monroeville, Pennsylvania, United States